CLINICAL TRIAL: NCT05757427
Title: Open-label,Single Site,Pilot Clinical Investigation to Assess Detectability and Sizing of Invasive Breast Cancers,Detectability of Benign Breast Lesions,Differentiation Between Malignant and Benign Breast Lesions Using Wavelia # 2
Brief Title: Pilot Clinical Evaluation of a Microwave Imaging System for Breast Cancer Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MVG Industries SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP.102.17.22.PAR
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will have an MBI scan with Wavelia in addition to standard of care procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients will have an MBI scan with Wavelia #2 in addition to standard reference imaging. (Experimental): Patients with an investigator assessed discrete breast abnormality of size >1cm and who attend the symptomatic breast unit for assessment as per standard of care protocol will be considered for participation in this clinical investigation.
  Interventions: Device: Wavelia #2

INTERVENTIONS:
Device: Wavelia #2 — Patients who are eligible and consent to have an MBI breast scan procedure will be asked to confirm their willingness to participate on the day of the breast scan. The patient will first have an Optical Breast Contour Detection (OBCD) scan, to reconstruct the external surface of the breast with high-precision, measure the total volume and the vertical extent of the breast before the MBI scan. The MBI scan will be performed on both breasts. The process will include optimization of breast positioning and breast cleaning to remove any transition liquid remaining on the skin.

SUMMARY:
The trialed investigational medical imaging device is a low-power microwave breast imaging system for cancer screening purposes. It is an active device which uses non-ionizing radiation.

Microwave imaging is an emerging imaging modality for the early detection of breast cancer. The physical basis of microwave imaging is the dielectric contrast between healthy and cancerous breast tissues at the microwave frequency spectrum.

This study is a pilot Clinical Evaluation of a microwave imaging system (Wavelia #2) for Breast Cancer Detection. The clinical data that will be collected in the context of this study is intended for the assessment of the imaging diagnostic capability and the safety of the investigational device.

DETAILED DESCRIPTION:
This study aims to enrol approximately 103 subjects presenting to the symptomatic breast unit with a breast abnormality who consent to undergo an Microwave Breast Imaging (MWBI) scan using the Wavelia #2 imaging system. The study uses an adaptive design to verify and validate the technical evolutions that have been integrated in the Wavelia# 2 prototype on a small patient dataset (30 patients). Once the technical performance has been established recruitment will continue to assess the clinical performance of the MBI system compared to standard of care reference imaging. The primary objectives of the study are to assess the performance of Wavelia # 2 in the detection of malignant and benign breast lesions, the sizing of malignant lesions for which post-surgery histology data will be available and the differentiation between benign and malignant breast abnormalities by means of features extracted from the MBI images.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Female subjects with an investigator assessed discrete breast abnormality of size > 1cm
* Able and willing to comply with the requirements of this study protocol
* Negative urine pregnancy test on the day of microwave imaging procedure (if of childbearing potential)
* intact breast skin (i.e., without bleeding lesion, no evidence of inflammation and/or erythema of the breast)
* Able to comfortably lie reasonably still in a prone position for approximately 15 minutes
* Have had biopsy more than 2 weeks prior to the microwave breast investigation (if applicable)

Exclusion Criteria:

* Have a cup size of A or whose breast is deemed too small to allow MBI assessment in the opinion of the investigator
* Are pregnant or breast-feeding
* Have had surgery on either breast within the past 12 months
* Have any active or metallic implant other than a biopsy clip
* Would be unsuitable for an MBI scan or unlikely to follow the protocol in the opinion of the Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kerin, Principal Investigator — Galway University Hospital
Locations (1):
- Galway University Hospital/Symptomatic Breast Unit, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All female patients with an investigator assessed discrete breast abnormality of size >1cm and who were called to attend the symptomatic breast unit for assessment as per standard of care protocol were considered for participation in this clinical investigation. If eligibility was confirmed patients were enrolled into the study and were scheduled for an MWBI either before or after standard of care assessments
Groups:
- Wavelia MWBI scan: Female patients who met all inclusion and exclusion criteria and completed an MWBI on both breasts with the technically validated MWBI
Period: Overall Study
Arm/Group | Wavelia MWBI scan
Started | 73
Completed | 62
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Device deficiency | 1
Not completed — All cysts aspirated before Wavelia scan | 1
Not completed — MWBI scan of only 1 breast | 3
Not completed — Invalid MWBI scan - various reasons - positioning, breast too large, patient movement | 5

BASELINE CHARACTERISTICS:
Population: Female patients who met all inclusion and exclusion criteria and completed an MWBI on both breasts with the technically validated MWBI
Arm/Group | Wavelia MWBI Scan
Number analyzed (Participants) | 62
Age, Customized [Median (Full Range); unit: years]
  Overall Demographics | 44 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Irish | 59
  Race/Ethnicity: Brazilian | 1
  Race/Ethnicity: Mauritian - South Asian | 1
  Race/Ethnicity: Romanian | 1
Region of Enrollment [Number; unit: participants]
  Ireland | 62

OUTCOME MEASURES:

1. Primary Outcome: Assess the Detectability Rate of Malignant and Benign Breast Lesions.
Description: Endpoint: Percentage of malignant and benign breast lesions correctly detected with Wavelia MWBI
Time Frame: 21 days
Population: Female patients who had a dominant discrete lesion in one breast who had a technically validated MWBI scan
Measure: Count of Units; unit: Dominant Lesions - Malignant & Benign
Units Other Than Participants: Dominant Lesions - Malignant & Benign
Arm/Group | Wavelia MWBI scan
Number analyzed (Participants) | 62
Number analyzed (Dominant Lesions - Malignant & Benign) | 62
Dominant Lesions - Malignant & Benign | 56
Statistical Analysis 1: Comparison: Wavelia MWBI scan; Test type: Other — The sample size is calculated solely for the first primary endpoint, no minimal number of benign nor malignant lesions was set. The sample size is calculated for this trial design, assuming a p1 = 75% and p0 = 60% for power (1-beta) of 80%, and an alpha level of 5%. We will conclude that the Wavelia # 2 Microwave Breast Imaging system is effective in detecting breast lesions if more than 43 of the 62 subjects' lesions are detected; Proportion of detected lesions = 90.32, 95% CI 2-sided [80.45 to 95.49]

2. Secondary Outcome: Correct Sizing of Breast Lesions With Wavelia MWBI
Description: Endpoint: Maximal linear size difference (in mm) between the MWBI lesion detection and the maximal size reported in the ultrasound lesion size estimates. This is measured as a continuous variable of difference in mm
Time Frame: 21 days
Population: Female patients for whom MWBI lesion size and Ultrasound lesion size data were obtained
Measure: Median (Full Range); unit: mm
Units Other Than Participants: All Lesions - Malignant & Benign
Arm/Group | Wavelia MWBI scan
Number analyzed (Participants) | 62
Number analyzed (All Lesions - Malignant & Benign) | 57
mm | -1.6 [-67.7 to 21.6]

3. Other Pre Specified Outcome: Evaluate the Wavelia MWBI Breast Lesion Detectability Rate on Patients With no Biopsy Clip
Description: Endpoint: Percentage of breast lesions correctly detected with Wavelia MWBI on patients with no biopsy clip marking in their breast
Time Frame: 21 days
Population: Female patients who did not have a biopsy clip in situ at time of MWBI scan
Measure: Count of Participants; unit: Participants
Arm/Group | Wavelia MWBI scan
Number analyzed (Participants) | 17
Participants | 15
Statistical Analysis 1: Comparison: Wavelia MWBI scan; Test type: Other — The percentage of malignant and benign breast lesions correctly detected by Wavelia MWBI on patients that did not have a biopsy clip marking the lesion position in the breast, will be presented with 95% confidence interval; Proportion of detected lesions = 88.24, 95% CI 2-sided [65.66 to 96.71]

4. Other Pre Specified Outcome: Safety Objective: Provide Further Data to Support the Establishment of the Safety Profile of MWBI Scan
Description: Endpoint: Incidence of Serious Adverse Events and Serious Adverse Device Effects during the total duration of the trial as well as other adverse events reported.
Time Frame: 21 days
Population: Female patients who consented to participate and had a complete or partial MWBI scan of at least one breast
Measure: Count of Participants; unit: Participants
Arm/Group | Wavelia MWBI scan
Number analyzed (Participants) | 73
Participants | 4
Statistical Analysis 1: Comparison: Wavelia MWBI scan; Test type: Other; Proportion of patients with AEs = 5.48

ADVERSE EVENTS:
Time Frame: 21 days
Description: Adverse Events and Adverse Device Effects were recorded from patient consent until the End of Study Follow Up Visit (up to 21 days post MWBI or prior to surgery, whichever happened first). Comprehensive assessments of any adverse event/device experienced by the subject was performed throughout the course of the study. Adverse events which occurred in Users or Other Persons (not study subjects) were also collected throughout the study along with device deficiencies
Arm/Group | Wavelia MWBI scan
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 4/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wavelia MWBI scan (N=73)
Immune system disorders (Immune system disorders) | 1 (1) — Allergic contact dermatitis
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck pain
General disorders and administration site conditions (General disorders) | 2 (2) — Chest discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT05757427/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT05757427/SAP_001.pdf